CLINICAL TRIAL: NCT05066867
Title: Compliance With Long-term Low-molecular-weight Heparin Prophylaxis/Treatment in the Anatenatal and Postnatal Population
Brief Title: LMWH Compliance in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cork University Maternity Hospital (Other)
Collaborators: HealthBeacon ICMS (Unknown)
Responsible Party: Principal Investigator, John R Higgins, Professor/Clinical Director, Cork University Maternity Hospital
Other Study IDs: CorkUMH
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Venous Thromboembolism; Antenatal Deep Vein Thrombosis
Keywords: Pregnancy thromboprophylaxis; LMWH compliance
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Smart sharps bin - collects data on compliance — collects compliance data

SUMMARY:
This is a prospective chart study that will aim to assess objective data on compliance levels to low molecular weight heparin (LMWH) injections among pregnant and postnatal women undergoing VTE thromboprophylaxis treatment at Cork University Maternity Hospital. This is a study that will help shine light on accurate data for compliance and possible factors affecting it, which will be useful for more individualised treatment plans for future patients. Patients at higher risk of Venous thromboembolism undergoing VTE thromboprophylaxis will be invited to participate in the study. Once the patient reads the information leaflet and signs consent, data will then be collected from the patients medical record. The patient will be given a smart sharps bin with an individual, unique product code. This device will be provided by HealthBeacon, a Dublin based start-up company. The device will be personalised with the treatment schedule pre-loaded onto it. When a used LMWH injection is disposed into the smart sharps bin, an infrared sensor is activated. The system captures an image of the injection in the chamber before moving it to the normal 'sharps' container of the bin for disposal. The captured image is time-stamped and sent to HealthBeacon's electronic database. HealthBeacon will only have the data pertaining to the disposal of injections for each sharps bin (i.e. the timing of the disposal of each used injection in each pre-coded bin). We are blinded to the compliance information and will only will receive the raw Data once treatment is completed. Data will be analysed to determine compliance of LMWH injections. This study will enable us to have a better insight on accurate compliance rates for LMWH injections in pregnant women at higher risk for venous thromboembolism (VTE). Understanding compliance with LMWH injections and the factors which can affect it, will hopefully guide future information and education that we offer to patients who are prescribed LMWH injections and help decrease maternal mortality rates in future.

ELIGIBILITY:
Inclusion Criteria:

* current VTE
* previous history of VTE
* class III obesity
* history of placenta mediated complications
* pre-eclampsia
* Advanced Maternal Age
* inherited thrombophilia
* prolonged immobilization
* varicose veins
* other risk factors that predispose them to VTE

Exclusion Criteria:

* life-long anti-coagulation
* mechanical heart valves
* other forms of injectable therapy for other illnesses
* long-term severe physical disability affecting mobility (eg: paraplegia, paralysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Antenatal and postnatal woman at higher risk of VTE commenced on LMWH thromboprophylaxis fitting the inclusion criteria
Study Population: Antenatal and postnatal women at higher risk of VTE, commenced on LMWH & fitting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
LMWH compliance levels in pregnancy | 18 months
  Compliance is described as a patient taking at least 80% of LMWH injections

SECONDARY OUTCOMES:
Sociodemographic factors | 18 months
  To determine sociodemographic factors that influence compliance

CONTACTS AND LOCATIONS:
Overall Officials: John RJ Higgins, M.D., Principal Investigator — CUMH
Locations (1):
- Cork University Maternity Hospital, Cork, Ireland